CLINICAL TRIAL: NCT02971657
Title: Bacterial Phenotype of Staphylococcus Aureus Has no Effect on Patients' Clinical Outcome in Orthopedic Device Related Bone Infections
Acronym: StaphType
Status: Completed | Type: Observational
Sponsor: BG Unfallklinik Murnau (Other)
Collaborators: AO Research Institute Davos (Other)
Responsible Party: Principal Investigator, Dr. Mario Morgenstern, MD, BG Unfallklinik Murnau
Other Study IDs: 2011-02
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Staphylococcal Infections
Keywords: Staphylococcus aureus phenotypic characterization; Antibiotic resistance; Orthopedic device related infections; Phenotypic characterization
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial samples from orthopaedic device related infections
Oversight: Data Monitoring Committee: No

SUMMARY:
This was a prospective study performed between November 2011 and September 2013. Patients with a confirmed S. aureus infection after fracture fixation or prosthetic joint infection were included. Exclusion criteria included infections involving external fixation pins, infections without any implanted hardware and culture positive patients not displaying any clinical sign of infection. The following surgical parameters were documented: affected bone or joint; type of implant; time between implantation of the device and onset of symptoms. Personal characteristics and patients'health status were also documented. Any revision surgeries involving the site of interest and all isolated pathogens were recorded throughout the course of treatment and follow-up.

A follow up examination was performed an average of 23 months after discharge. Primary outcome at follow up was cure. Cure was defined by the authors as: missing local (at site of interest) or systemic signs of infection, terminated surgical and systemic therapy and restoration of joint or limb function.

At the first surgical procedure after enrolment, at least four deep bone biopsies were taken from the interface between implant and affected bone. Identification and antibiotic susceptibility testing of all growth was performed. Multi-drug-resistance (MDR) was defined according to the definitions of the European Committee of Antimicrobial Susceptibility Testing (EUCAST). Biofilm formation was analysed and quantified in microtitre plate assays according to protocol of Stepanovic et al.(see references).

DETAILED DESCRIPTION:
This was a prospective study performed between November 2011 and September 2013. All patients provided informed written consent prior to inclusion in the study. Inclusion criteria were deep S. aureus infections after fracture fixation or prosthetic joint surgery. Fracture fixation infections includes fractures involving the long bones as well as the pelvis and the spine. Bacterial growth at the site of interest in combination with either pseudarthrosis, implant-loosening/failure or local and systemic signs of surgical site infection were required for inclusion. Exclusion criteria included infections involving external fixation pins, infections without any implanted hardware and culture positive patients not displaying any clinical sign of infection.

Upon entry into the study, the following surgical parameters were documented: affected bone or joint; type of implant; time between implantation of the device and onset of symptoms. Personal characteristics were also documented and included: gender; age; body mass index (BMI); smoker/non-smoker; overall medical condition (Charlson comorbidity index); and chronic immunosuppressive conditions (Diabetes mellitus, chronic alcoholism, Child's class C cirrhosis, neoplasia, transplantation, AIDS and steroid medication). Any revision surgeries involving the site of interest and all isolated pathogens were recorded throughout the course of treatment and follow-up.

A follow up examination was performed an average of 23 months after discharge. Primary outcome at follow up was cure. Cure was defined by the authors as: missing local (at site of interest) or systemic signs of infection and terminated surgical and systemic therapy.

At the first surgical procedure after enrolment, at least four deep bone biopsies were taken from the interface between implant and affected bone. The tissue samples were placed in a sterile container with thioglycollate liquid medium (bioMérieux, Hazelwood, MO, USA). The samples were cultured for ten days at 37°C and examined each day macroscopically. Any growth was inoculated onto a blood agar plate (bioMérieux, Hazelwood, MO, USA) for further growth and subsequent identification. In all cases, additional swabs and soft tissue samples may have been taken as per clinical routine, however, only samples adjacent to the implant were used for diagnosis in this study.

Identification and antibiotic susceptibility testing of all growth was performed using a Vitek2 (bioMerieux Vitek Inc, Hazelwood, MO, USA). Multi-drug-resistance (MDR) was defined according to the definitions of the European Committee of Antimicrobial Susceptibility Testing (EUCAST). Oxacillin resistance was used as an indicator for methicillin resistant S. aureus (MRSA).

Biofilm formation was analysed and quantified in microtitre plate assays according to the well-established protocol of Stepanovic et al.(see references).

The key variables with regards to bacterial phenotype were: biofilm formation; methicillin resistance;multidrug resistance;staphyloxanthin production and hemolysis. The primary outcome measure was whether the infection was "cured" or not. Primary outcome parameters were calculated as a function of all patients for whom data was complete. Statistical comparison was restricted to the lower extremity cohort since the other patients are not scored for many of the functional outcome measures and as such incomplete.

Univariate logistic regression models were used to determine the influence of each prognostic factor (obesity, smoking, diabetes mellitus, chronic immune suppression, open fracture (initially), early onset infection, biofilm formation, methicillin resistance, MDR and Charlson comorbidity index) on cure. P-values <0.05 were considered significant. Statistical analyses were performed using SAS software (Version 9.2; Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Infections after fracture fixation or prosthetic joint surgery
* Affected bone or joint: Long bones of the lower and upper extremity
* Bacterial growth of S. aureus at the site of interest
* Written consent
* Age: 18 and older

Exclusion Criteria:

* no prove of bacterial growth at site of interest
* missing consent
* infections involving external fixation pins, infections without any implanted hardware.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Orthopaedic device related infection involving longbones of the upper and lower extremities
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cure | 23 months
  Cure was defined by the authors as: missing local (at site of interest) or systemic signs of infection and terminated surgical and systemic antibiotic therapy. All Parameters had to be positive to fulfill the outcome parameter "cure".If one of the mentioned parameters was negative, outcome was defined as "not cured". Local signs of infection were defined as the appearance of: redness, tenderness, swelling or persisting wound drainage.

REFERENCES:
- [Background] Stepanovic S, Vukovic D, Hola V, Di Bonaventura G, Djukic S, Cirkovic I, Ruzicka F. Quantification of biofilm in microtiter plates: overview of testing conditions and practical recommendations for assessment of biofilm production by staphylococci. APMIS. 2007 Aug;115(8):891-9. doi: 10.1111/j.1600-0463.2007.apm_630.x. PMID 17696944
- [Background] Post V, Wahl P, Uckay I, Ochsner P, Zimmerli W, Corvec S, Loiez C, Richards RG, Moriarty TF. Phenotypic and genotypic characterisation of Staphylococcus aureus causing musculoskeletal infections. Int J Med Microbiol. 2014 Jul;304(5-6):565-76. doi: 10.1016/j.ijmm.2014.03.003. Epub 2014 Apr 3. PMID 24768432